CLINICAL TRIAL: NCT06268743
Title: Understanding the GUT Microbiome Through a Fitness Intervention of Aerobic and Resistance Training for Individuals With Type 2 Diabetes Mellitus (GUTFIT Study)
Brief Title: Effects of a Combined Exercise Intervention on the Gut Microbiome of People With Type 2 Diabetes
Acronym: GUTFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Martin Senechal, Full Professor, Martin Senechal, Ph.D., University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-114
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes
Keywords: Exercise intensity; Aerobic training; Resistance training; Gut microbiome; Physical activity; Glycemia; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Parallel group, single blinded, randomized trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity (Experimental): Participants will perform high-intensity aerobic and strength training exercises.
  Interventions: Other: High intensity
- Moderate Intensity (Active Comparator): Participants will perform moderate-intensity aerobic and strength training exercises.
  Interventions: Other: Moderate intensity

INTERVENTIONS:
Other: High intensity — High intensity exercise
  Arms: High intensity
Other: Moderate intensity — Moderate intensity exercise
  Arms: Moderate Intensity

SUMMARY:
The goal of this experimental trial is to learn about the changes in bacterial diversity in individuals with type 2 diabetes who perform endurance and strength training at different intensities.

Participants with type 2 diabetes will be randomly assigned to 16 weeks of either moderate-intensity endurance and strength training or high-intensity endurance and strength training.

Researchers will compare the moderate-intensity and high-intensity exercise groups for differences in glycemia and bacterial diversity.

DETAILED DESCRIPTION:
It is unclear if performing aerobic training (AT) and resistance training (RT) at a higher intensity in people with type 2 diabetes mellitus (T2DM) would generate greater improvement in HbA1c and if this would be associated with increased gut microbiome diversity.

Therefore, the objective of this study is to test whether performing resistance training and aerobic exercise (RT+AT) at a high intensity for 16 weeks will significantly improve glycemic control (HbA1c) and if this change is associated with an increase in gut microbiome diversity compared to performing RT+AT at a moderate intensity in individuals with poor glycemic control. We hypothesize that individuals performing RT+AT at a high intensity will significantly reduce HbA1c and improve gut microbiome diversity compared to individuals performing RT+AT at a moderate intensity.

Methods: This study is a parallel-group, single-blinded, randomized trial including 40 adults (50% males and females) living with T2DM. Participants will be allocated to one of two treatment groups: 1) high intensity or 2) moderate intensity for 16 weeks.

A total of 40 participants (n = 20 for each sex) living with T2DM with poor glycemic control (HbA1c => 7.0%), aged between 19-64 years, who do not currently meet the recommended levels of physical activity for optimal health, (i.e., 150 min of moderate-to-vigorous physical activity + 2 days/week of resistance training) will be recruited.

Intervention: Participants will undergo a supervised exercise intervention of RT+AT for 16 weeks, performed at high or moderate intensity. 1) High intensity: AT will be performed at 70-80% heart rate reserve and 8-10 repetitions (75-80% maximal strength). 2) Moderate intensity: AT will be performed at 45-55% heart rate reserve and 12-15 repetitions (65-70% maximal strength). AT will consist of expending 10 kcal/kg per week, while RT will consist of 2 days of resistance training per week as per the recommendations. Our previous work shows that participants could perform this type of intensity; therefore, no problems are anticipated. Exercise intensity will be monitored using heart rate for aerobic training and the OMNI-RES scale (1-10) for resistance training.

Primary Outcomes: All HbA1c tests will be performed using a validated DCA Vantage® Analyzer (Siemens, Germany). Participants will undergo HbA1c tests at baseline and post-intervention (16 weeks). The gut microbiome composition will be determined at baseline and post-intervention in participant feces using next-generation sequencing (Illumina MiSeq) of 16S ribosomal RNA genes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 - 64 years old;
* Diagnosed with type 2 diabetes;
* An HbA1c >= 7.0%;
* Not currently meeting the recommended levels of physical activity for optimal health (i.e., 150 minutes of moderate-to-vigorous physical activity and 2+ days/week of resistance training);
* Average less than 10,000 steps per day over the last seven days;
* No change in diabetes medications over the last three months.

Exclusion Criteria:

* Not diagnosed with type 2 diabetes;
* Partaking in a self-reported regular exercise regimen, defined as consistent participation in running or jogging activity, attending exercise classes every week, or averaging 10,000 steps per day or more over seven days;
* Currently performing two days of resistance training per week;
* Having an injury that would prevent safe participation in the intervention;
* A self-reported diagnosis of low iron concentrations, anemia, or being treated for these conditions;
* A diagnosis of any red blood cell altering condition (i.e., sickle cell anemia, poikilocytosis);
* Currently living with any cardiovascular disease which would impact the ability to participate in exercise safely;
* Currently prescribed any medication which would impact the ability to use a heart rate monitor to accurately track intensity.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Glycemic control through glycated hemoglobin | 16 weeks
  Change in glycated hemoglobin (HbA1c)
Gut microbiome diversity through 16S ribosomal RNA genes | 16 weeks
  Change in the composition of the gut microbiome based on sequencing of 16S ribosomal RNA genes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, Ph.D., Principal Investigator — University of New Brunswick
Locations (1):
- Cardiometabolic Exercise & Lifestyle Laboratory, Fredericton, New Brunswick, Canada